CLINICAL TRIAL: NCT04530253
Title: A Study on the Post-acute Care for Cardiovascular Disease
Brief Title: The Post-acute Care for Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22373
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: the Demands of Post-acute Care in Cardiovascular Disease
Keywords: Post-acute care; Cardiovascular disease; nursing; protocol
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim: The aims of this study are 1) to determine the demand of post-acute care among patients with cardiovascular disease in China; 2) to identify the details of demands especially which have value for the post-acute care for patients with cardiovascular disease.

Design: A single center prospective cohort study. Methods: Patients will be enrolled from the department of cardiology in a tertiary teaching hospital. The data on the demands of post-acute care will be collected throughout the hospitalization and discharge. Patients with cardiovascular disease will be followed up for 3 months. The study was approved by the ethics committee in August 2020.

Discussion: Post-acute care is very important for the short- and long-term outcomes of the patients with cardiovascular disease. This study will provide an effective tool for the investigation of the detailed demands for post-acute care in cardiovascular disease and provide a better understanding of the demands for the patients with cardiovascular disease.

Impact: In clinical practice, understanding of the demands for post-acute care of the patients with cardiovascular disease can help nurses implement effective strategies at the early stages to patients to improve the short- and long-term outcomes of the patients. The follow-up results will help us better understand the impact of a post-acute care system on patients' outcomes.

Keywords: Post-acute care, Cardiovascular disease, nursing, protocol

DETAILED DESCRIPTION:
1. INTRODUCTION China has entered the high-pressure period of cardiovascular disease. The incidence of cardiovascular disease is still rising. It has become a great threaten for the health of Chinese resident and the social economy development. The comprehensiveness and complexity of the influencing factors of cardiovascular disease determine the long-term and arduous task of prevention and treatment. It is necessary to coordinate the resources of all parties and improve the mechanism of comprehensive prevention and treatment of cardiovascular disease with multi department cooperation. At present, due to the limited medical resources, high cost of hospitalization and the shortage of hospital beds, the average length of stay of patients is gradually shortened, resulting in an increasing number of patients with cardiovascular disease who are discharged immediately after acute treatment. Although the emergency problems of the disease have been solved during hospitalization, there is still a period of transition in the process of rehabilitation before returning to the family and society. Therefore, long-term and systematic management after discharge is the most important measure to improve the prognosis of patients with cardiovascular disease. Post-acute care (PAC) is the most important guarantee to provide continuous medical care for patients with cardiovascular diseases. Readiness for hospital discharge is the key link between emergency care and post-acute care, which helps to shorten the length of hospital stay, reduce the rate of readmission, improve the quality of life of patients with cardiovascular diseases and reduce medical costs. In recent years, China's post-acute care system has made a series of achievements, but it is still distributed in the form of dots, and there is no mature working mode. Therefore, it is urgent to build a characteristic post-acute care system for cardiovascular diseases based on China's national conditions. However, Understanding the details of patients' demands is the key and the first step in building the post-acute care system for cardiovascular diseases. This study will provide an effective tool for the investigation of the detailed demands for post-acute care in cardiovascular disease and provide a better understanding of the demands for the patients with cardiovascular disease.
2. THE STUDY 2.1 Aims The aims of this study are 1) to determine the demand of post-acute care among patients with cardiovascular disease in China; 2) to identify the details of demands especially which have value for the post-acute care for patients with cardiovascular disease.

2.2 Study Design This is a single-center, prospective cohort study conducted at a tertiary teaching hospital in Shanghai, China.

2.3 Setting The study will be conducted in the cardiology department in Zhongshan hospital, Shanghai, China, which is the largest hospital in Shanghai with 2005 beds.

Cardiology department focuses on interventional diagnosis and treatment of complex and difficult cardiovascular diseases with 527 beds and 503 nurses and physicians. Approximately more than 24000 patients per year are admitted, including angina pectoris, acute myocardial infarction, atrial fibrillation, atrial flutter, premature ventricular contractions, atrioventricular block, sick sinus syndrome, pulmonary hypertension, congenital heart disease, rheumatic heart disease, valvular disease, heart failure, cardiomyopathy, myocarditis, etc.

2.4 Participants Inclusion Criteria Patients with cardiovascular disease aged above 18. The patients are aware of the disease condition. The patients can read and understand independently and participate in this study voluntarily.

Exclusion Criteria The patient's condition is critical and life-threatening. People who are not conscious or are not cooperative by mental disorders. Patients refused to continue to participate in the study.

2.5 Sample size Our study will aim to identify demands for the post-acute care of patients with cardiovascular disease. According to the rule of thumb, the sample size should be 5-10 times the number of items of questionnaire. Considering the 20% loss rate, the sample size is required to be at least 900 cases, and 1000 cases are preliminarily planned to be included in our hospital.

2.6 Data collection Demands for post-acute care Data of the demands for post-acute care will be collected face to face or telephone, including guidance of rehabilitation exercise, medication, diet, introduction of available social resources support, such as long-term care insurance, etc. Demographic characteristic The demographic variables and related information on the demands of post-acute care will also be collected, including gender, age, marital status, education level, work status, family per capita monthly income, type of medical insurance, distance between home and hospital, main diagnosis, duration of illness, pipeline indwelling, length of hospital stay, hospitalization treatment, medication, the destination after discharge, etc.

Readiness for hospital discharge scale (RHDS) The original scale was developed by Weis et al. It has 4 dimensions: self-condition, disease knowledge, coping ability after discharge, social support available, and 23 items. The first question is not included in the total score. The rest items are scored by 0-10 points. The score of "0" represents "not knowing at all" and "completely unable", and "10" stands for "completely knowing" and "completely capable". Patients can choose the appropriate score according to their own situation. The higher the score, the better the readiness for discharge. This study adopts the Chinese version of Zhao et al. of West China Hospital of Sichuan University.

2.7 Data management All the data will be entered and stored in the Research Electronic Data Capture (REDCap), which will be securely locked, and password protected. It is supported and maintained by the Evidence-based center of Fudan University. Data management and analysis, including data audit, import and tracking will be done by the biostatisticians in the center. Each patient will be given a study identification number; all paper files will be imported to the database once completed.

2.8 Statistical analysis Chi square test was used for categorical data, t-test and ANOVA were used for measurement data. Through univariate, multivariate analysis, structural equation model and path analysis, the relationship between readiness for hospital discharge and demands of patients for post-acute care was analyzed.

2.9 Ethical considerations This study was approved by the Hospital Ethics Board in August 2020 (SK2020-014). The study will be conducted in accordance with the International Council for Harmonization and Good Clinical Practice principles. The study will adhere to the ethical principles stated in the Declaration of Helsinki.

All patients will receive written and verbal information of the study before surgery. Written informed consent will be obtained before inclusion. Patient have the right to withdraw from the study at any time. Data collection will be stopped, and patients' record will be deleted from the database if a patient withdraws from the study.

2.10 Validity, reliability and rigor In this study, we will use one instrument named RHDS. The validity and reliability will be tested with the baseline data. The cohort study will follow the STROBE statement.

ELIGIBILITY:
Inclusion Criteria:

Patients with cardiovascular disease aged above 18. The patients are aware of the disease condition. The patients can read and understand independently and participate in this study voluntarily.

Exclusion Criteria:

The patient's condition is critical and life-threatening. People who are not conscious or are not cooperative by mental disorders. Patients refused to continue to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the cardiology department in Zhongshan hospital, Shanghai, China. Patients with cardiovascular disease will be included
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Demands for post-acute care | 2020/10/1~2022/9/30
  The demands for post-acute care will be collected face to face or telephone, including guidance of rehabilitation exercise, medication, diet, introduction of available social resources support, such as long-term care insurance, etc.
Readiness for hospital discharge scale (RHDS) | 2020/10/1~2022/9/30
  It has 4 dimensions: self-condition, disease knowledge, coping ability after discharge, social support available, and 23 items.

IPD SHARING:
Plan to Share IPD: No